CLINICAL TRIAL: NCT04903821
Title: Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Elinzanetant in Participants With Impaired Hepatic Function (Classified as Child-Pugh A or B) in Comparison to Matched Controls With Normal Hepatic Function.
Brief Title: A Study to Learn How Different Levels of Decreased Liver Function Influence Blood Levels of Elinzanetant Compared to Normal Liver Function in Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21668; 2020-005939-74 (EudraCT Number)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Child- Pugh A) (Experimental): Participants with mild impaired hepatic function (Child-Pugh A), including at least 2 female participants.
  Interventions: Drug: BAY3427080
- Group B (Child-Pugh B) (Experimental): Participants with moderate impaired hepatic function (Child-Pugh B), including at least 2 female participants
  Interventions: Drug: BAY3427080
- Control A match controls for group A (Experimental): Matched control participants for Group A with normal hepatic function.
  Interventions: Drug: BAY3427080
- Control B match controls for group B (Experimental): Matched control participants for Group B with normal hepatic function
  Interventions: Drug: BAY3427080

INTERVENTIONS:
Drug: BAY3427080 — Orally administered, single dose on Day 1 and single does once daily on Day 3 to 8

SUMMARY:
Researchers are looking for a better way to treat people who have symptoms caused by hormonal changes, like those that happen in women during menopause. These symptoms can include vasomotor symptoms. Before a treatment can be approved for patients to take, researchers do clinical studies to better understand its safety and what happens to the treatment in the body.

The study drug, elinzanetant, was designed to treat vasomotor symptoms. The liver plays an important role in removing elinzanetant from the body. Therefore, this study is done to find out how reduced liver function influences the removal of elinzanetant.

The study will include male and female participants who are 18 to 75 years old. One part of the participants will have mildly or moderately impaired hepatic function. For each group with impaired hepatic function, a group with normal hepatic function will be included.

Blood and urine samples will be collected. The physician will also check the participants' heart health using an electrocardiogram (ECG). The participants will answer questions about their well-being and taken medications.

The researchers will compare the blood levels of elinzanetant in the participants with impaired hepatic function to those of the matched participants with normal hepatic function. This way, they can see how blood levels of elinzanetant are influenced by liver function. This information is important for giving recommendations on dosing in patients with impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
* Participants who have

  * Impaired hepatic function according to Child-Pugh score A or B,
  * Documented medical history of liver cirrhosis confirmed by either histopathology, laparoscopy, fibroscan, computer tomography, magnetic resonance imaging (MRI), or ultrasound,
  * Stable impairment for at least 2 months prior to screening in the judgment of the investigator.
* Participants who have normal hepatic function and are overtly healthy.
* Body weight of at least 50 kg and BMI within the range 18 to 38 kg/m*2 (inclusive).
* Male or female Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Male participants:

    * Male participants of reproductive potential must agree to use a condom (with or without spermicide) when heterosexually active. This applies for the time period between the signing of the informed consent form (ICF) until 7 days after the last dose of study intervention.
    * Female partners of male participants do not need to follow special precautions.
  * Female participants of childbearing potential: have to agree to use a highly effective non-hormonal contraception when heterosexually active. This applies for the time between signing the ICF until 21 days after the last dose of study intervention (for details and definitions of childbearing potential and allowed contraceptive methods).
* Female participants of childbearing potential must have a negative pregnancy test at screening and on Day -1.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Ascites qualitatively estimated as severe or requiring acute or frequent paracentesis.
* Renal failure with an estimated glomerular filtration rate (eGFR) <= 40 mL/min according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Encephalopathy of > grade 2.
* Renal failure with an eGFR <=60 mL/min CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation.
* Any clinically relevant disease (other than those related to hepatic impairment for the hepatic impaired participants) within 4 weeks prior to study drug administration including.
* Medically relevant infections and acute gastro-intestinal diseases (vomiting, diarrhea, constipation).
* Severe cerebrovascular or cardiovascular disorders less than 6 months prior to dosing, e.g., stroke, myocardial infarction, unstable angina pectoris, congestive heart failure of grade III or IV according to New York Heart Association (NYHA), arrhythmia requiring antiarrhythmic treatment, percutaneous transluminal coronary angioplasty or coronary artery bypass graft.
* Febrile illness within 1 week before first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Cmax,md,u of elinzanetant | On day 8
  Cmax,md,u: Maximum observed drug concentration in measured matrix after multiple dose administration during a dosage interval of the unbound analyte.
AUC(0-24)md,u of elinzanetant | On day 8
  AUC: Area under the curve extrapolated to infinity. AUC(0-24)md,u: AUC from time 0 to 24 after multiple dosing of the unbound analyte.

SECONDARY OUTCOMES:
Incidence of treatmentemergent adverse events (TEAEs) | About 10 months
Severity of treatmentemergent adverse events (TEAEs) | About 10 months
AUCu of elinzanetant | On Day 1
  Or AUC(0-tlast) if AUC cannot be determined. AUCu: AUC extrapolated to infinity of the unbound analyte. AUC(0-tlast): AUC from time 0 to the last data point > LLOQ (lower limit of quantification)
Cmax,u of elinzanetant | On Day 1
  Cmax,u: Maximum observed drug concentration in measured matrix after single dose administration of the unbound analyte.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - APEX GmbH, München, Bavaria
  - CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.